CLINICAL TRIAL: NCT03268161
Title: Observational Study of the Prevalence of Some Genetic Mutations in Patients With Neuropathy Associated With Anti-Myelin-associated Glycoprotein (MAG) Antibodies.
Brief Title: Prevalence of Genetic Mutations in Patients With Neuropathy Associated With Anti-Myelin-associated Glycoprotein (MAG) Antibodies
Acronym: GENOMAG
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_3018
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Neuropathy Demyelinating
Keywords: anti-MAG neuropathy; Waldenström disease; Mutational analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Medullary or blood sample stored in a bio-bank during lymphocyte phenotyping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with anti-MAG neuropathy: Mutational analysis of clonal B cells
  Interventions: Diagnostic Test: Mutational analysis of clonal B cells

INTERVENTIONS:
Diagnostic Test: Mutational analysis of clonal B cells — Mutational analysis based on medullary or blood samples stored in a bio-bank during routine lymphocyte phenotyping.
  Mutations affecting MYD88 (MYD88 L265P mutation), CXCR4 (Whim-like CXCR4 mutation) loci are sought.

SUMMARY:
Anti-MAG (Myelin Associated Glycoprotein) neuropathy is related to clonal B lymphocyte proliferation producing an monoclonal immunoglobulin (IgM) with anti-MAG activity. IgM may be a reflection of malignant lymphoproliferative syndrome (Waldenström disease) or, more often, monoclonal gammopathy of unknown significance.

The anti-MAG antibody has a direct toxicity on the myelin sheath of the peripheral nervous system responsible for a length-dependent demyelinating polyneuropathy. Clinically, this results in a sensitive, ataxic predominant polyneuropathy in the lower limbs, sometimes associated with a tremor of attitude and action tremor of the upper limbs.

Clonal B cells at the origin of IgM production may have acquired mutations affecting MYD88 (MYD88 L265P mutation) and CXCR4 (Whim-like CXCR4 mutation). The prevalence of the MYD88 L265P mutation is estimated to be 50% in monoclonal gammopathies of undetermined significance and more than 80% in Waldenström disease. CXCR4 Whim-like mutations are found in 40% of patients with Waldenström's disease.

No studies have reported the prevalence of these mutations in patients with anti-MAG neuropathies.

DETAILED DESCRIPTION:
This is a retrospective observational study in patients with anti-MAG neuropathy. Mutational analysis will be performed for patients with a medullary or blood sample stored in a bio-bank during lymphocyte phenotyping. This phenotyping was carried out most often in search of a malignant haemopathy associated with the monoclonal peak. No new samples were taken from the patient (blood or spinal cord).

Immunoglobulin gene rearrangement of the clonal B cells are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anti-MAG neuropathy
* Blood and/or bone marrow samples available in bio-bank
* Given informed consent

Exclusion criterion

* Participation refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anti-MAG neuropathy followed in the Internal Medicine Ward of the Rennes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of MYD88 L265P mutations in anti-MAG neuropathies | At inclusion : after the patient's given consent
  Mutational status of MYD88 L265P is assessed using high-throughput sequencing (HTS) and allele specific polymerase chain reaction (AS-PCR)
Prevalence of CXCR4 Whim-like mutations in anti-MAG neuropathies | At inclusion : after the patient's given consent
  Mutational status of CXCR4 is assessed using HTS and AS-PCR

SECONDARY OUTCOMES:
Immunoglobulin gene rearrangement | At inclusion : after the patient's given consent
  Immunoglobulin gene rearrangements are determined with a multiplex PCR

CONTACTS AND LOCATIONS:
Overall Officials: Olivier DECAUX, MD, PhD, Study Director — CHU Rennes
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No